CLINICAL TRIAL: NCT02086799
Title: Is There a Role for Thyroid Hormones Treatment in the Set-up of Acute Moderate to Severe Asthma Exacerbation
Brief Title: Thyroid Hormones Treatment in Asthma Exacerbation
Acronym: THINAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 354-13CTIL
Record Dates: First submitted 2014-02-11; First posted 2014-03-13 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Asthma
Keywords: asthma; thyroid hormones; treatment; asthma exacerbation
MeSH Terms: conditions — Asthma | interventions — Thyroxine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV thyroxin (Experimental): IV thyroxin
  Interventions: Drug: IV thyroxin
- control IV saline (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IV thyroxin — Patients will receive treatment with intra-venous thyroxine 100mcg once on admission and additional 100mcg after 12 hours.
  Other Names: elthyroxin; thyroxin; euthrux
  Arms: IV thyroxin
Drug: Placebo — Patients will receive treatment with normal saline 100ml once on admission and additional 100ml after 12 hours
  Other Names: saline
  Arms: control IV saline

SUMMARY:
This study will explore whether supplementation with thyroid hormones in the set-up of asthma exacerbation could improve the clinical outcomes.

The study will include adults admitted to Rambam health care campus for moderate to severe Asthma exacerbation.

The study is a prospective, randomized, double-blind, placebo-controlled, clinical trial. Patients will be randomized on admission to receive treatment with intra-venous thyroxine (100mcg once on admission and additional 100mcg after 12 hours) or placebo. The study treatment will be given only after the initial bronchodilator therapy, oxygen and informed consent are given. The primary endpoint is the time to return of the peak expiratory flow (PEF) rate to normal values or personal base line.

DETAILED DESCRIPTION:
Study population: The study will include adults admitted to Internal Medicine B (IMB) department, Internal Medicine H (IMH) department or medical intensive care unit (MICU) in Rambam-Health Care Campus for moderate to severe Asthma exacerbation. The severity of the exacerbation will be based on several acceptable clinical and laboratory criteria, including breathless, alertness, pulse rate, respiratory rate, partial pressure of oxygen in arterial blood (PaO2), partial pressure of carbon dioxide in arterial blood (PaCO2), oxygen saturation, peak expiratory flow (PEF). Study protocol: The study is a prospective, randomized, double-blind, placebo-controlled, clinical trial. Patients will be randomized on admission to receive treatment with intra-venous thyroxine (100mcg once on admission and additional 100mcg after 12 hours) or placebo. The study treatment will be given only after the initial bronchodilator therapy, oxygen and informed consent are given. The primary endpoint is the time to return of the PEF rate to normal values or personal base line. PEF rates will be examined first after initial bronchodilator therapy and then, every 8 hours.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Known Asthma
* The exacerbation is defined as moderate or severe.
* Not currently enrolled as an active participant in another clinical trial of a medical therapy or device.
* The patient or first degree family relative (in cases where the patient is intubated) has authorized his/her consent to participate in this trial. The patient will be asked to give his consent only after initial bronchodilator therapy

Exclusion Criteria:

* 60 years of age or older
* Known thyroid disorders
* Subject where thyrotoxicosis is suspected
* Known heart disease
* Heart rate > 140

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
time to normalization of PEF (peak expiratory flow) | one week
  The primary endpoint is the time to return of the PEF rate to normal values or personal base line.

SECONDARY OUTCOMES:
Length of stay | one week
  • Length of stay (in cases of hospitalization in the internal medicine departments) or length of intubation (in cases of hospitalization in the MICU).
Time to oxygenation | one week
  Time to oxygen saturation > 95% (while breathing spontaneously and without oxygen supplements)
heart rate | one week
  Time to normalization of heart rate
respiratory rate | one week
  Time to normalization of respiratory rate

CONTACTS AND LOCATIONS:
Overall Officials: Zaher S Azzam, prof., Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam health care campus, Haifa, Israel